CLINICAL TRIAL: NCT06535204
Title: Effects of Oral Administration of Anthriscus Sylvestris Leaves on Mild Knee Osteoarthritis: A Randomized, Double-Blind, Placebo-Controlled Clinical Trial
Brief Title: Effects of Anthriscus Sylvestris Leaves on Mild Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pusan National University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: H-1905-043-079
Record Dates: First submitted 2024-07-14; First posted 2024-08-02 (Actual); Last update posted 2024-08-02 (Actual); Status verified 2024-07

CONDITIONS: Osteoarthritis; Articular Cartilage; Functional Food
MeSH Terms: conditions — Osteoarthritis | interventions — microcrystalline cellulose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): The intervention group consumed the test food twice daily (400 mg in the morning and 400 mg in the evening, each time as one hard capsule), 30 minutes after eating, with water. The administration period lasted 12 weeks for each participant.
  The test food is named Aqueous extract of A. sylvestris leaves. The ingredients and their contents are as follows: Aqueous extract of A. sylvestris leaves 62.5%, Microcrystalline Cellulose 35.5%, Silicon Dioxide 1.0%, Magnesium Stearate 1.0%. The dosage form is a hard capsule, with a content weight of 400 mg per capsule.
  Interventions: Dietary Supplement: Aqueous extract of A. sylvestris leaves
- Control Group (Placebo Comparator): The Control group consumed the test food twice daily (400 mg in the morning and 400 mg in the evening, each time as one hard capsule), 30 minutes after eating, with water. The administration period lasted 12 weeks for each participant.
  The test food is named Microcrystalline Cellulose. The ingredients and their contents are as follows: Microcrystalline Cellulose 98%, Silicon dioxide 1.0%, Magnesium stearate 1.0%. The dosage form is a hard capsule, with a content weight of 400 mg per capsule.
  Interventions: Dietary Supplement: microcrystalline cellulose

INTERVENTIONS:
Dietary Supplement: Aqueous extract of A. sylvestris leaves — Provided functional food made from Aqueous extract of A. sylvestris leaves
  Arms: Experimental Group
Dietary Supplement: microcrystalline cellulose — Provided placebo composed of microcrystalline cellulose instead of A. sylvestris leaf extract.
  Arms: Control Group

SUMMARY:
Osteoarthritis (OA) is a common degenerative joint disorder that causes pain, stiffness, and functional impairment. Current treatments for OA are limited to symptom relief and have potential side effects. Anthriscus sylvestris leaves are a natural remedy that has been shown to have anti-inflammatory and cartilage-protective effects in animal models of OA.

DETAILED DESCRIPTION:
Osteoarthritis (OA) is a common degenerative joint disorder that causes pain, stiffness, and functional impairment. Current treatments for OA are limited to symptom relief and have potential side effects. Anthriscus sylvestris leaves are a natural remedy that has been shown to have anti-inflammatory and cartilage-protective effects in animal models of OA. A randomized, double-blind, placebo-controlled trial was conducted with 100 participants aged 40 to 75 with Kellgren & Lawrence grade 1 or 2 knee OA. Participants were assigned to receive either 500 mg of Anthriscus sylvestris leaves extract or placebo daily for 12 weeks. The primary outcome was the change in the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) score from baseline to week 12. Secondary outcomes included the changes in visual analogue scale (VAS) for pain, C-reactive protein (CRP), and erythrocyte sedimentation rate (ESR) from baseline to week 12. The Anthriscus sylvestris leaves extract group showed a significant improvement in the total WOMAC score, as well as the pain, stiffness, and physical function sub-scores, compared with the placebo group after 12 weeks of treatment. The Anthriscus sylvestris leaves extract group also showed a significant reduction in VAS and CRP, but not in ESR, compared with the placebo group. No adverse events or safety concerns were reported in either group. Anthriscus sylvestris leaves extract enhanced joint and cartilage health in humans with mild OA symptoms, as indicated by the reduction in WOMAC, VAS, and CRP. The extract was also safe and well-tolerated. Anthriscus sylvestris leaves extract may be a promising natural alternative for the management and prevention of OA.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 40 to 75 years, regardless of gender
* Individuals with a Visual Analogue Scale (VAS) score of 3/10 or higher
* Individuals with a Kellgren & Lawrence grading scale of grade 1 or 2, determined by 'Both Knee Joint AP/LAT' radiographs
* Individuals who have had a washout period of at least 4 weeks for arthritis- related medications or health supplements
* Individuals capable of normal physical activity who have voluntarily provided written informed consent to participate in this study

Exclusion Criteria:

* Individuals with a history of fractures within the past year
* Individuals with osteophytes around the joints, irregular joint surfaces, or subchondral bone cysts, indicating moderate arthritis
* Individuals currently undergoing treatment for a diagnosed thyroid disorder
* Individuals with kidney disease or serum creatinine levels of 1.4 mg/dL or higher
* Individuals with proteinuria of 2+ or higher
* Individuals with liver disease or AST or ALT levels of 100 IU/L or higher
* Individuals with uncontrolled hypertension or heart conditions such as angina or myocardial infarction
* Individuals taking medication for psychiatric disorders, except for intermittent medication for sleep disorders
* Individuals who have taken herbal or medicinal decoctions within the past two months
* Individuals who have received other investigational drugs within the past four weeks
* Individuals who need to continuously take medication that may affect the outcome of the study
* Individuals with a history of gastrointestinal resection surgery (excluding appendectomy)
* Pregnant or breastfeeding women
* Individuals with alcoholism or those who drink more than four times per week regularly
* Individuals with hypersensitivity to the test food or its ingredients
* Individuals who may be uncooperative or deemed incapable of completing the study by the investigator
* Individuals with arthritis due to specific factors other than degeneration, as determined by the principal investigator

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2019-06-24 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2020-04-30 (Actual)

PRIMARY OUTCOMES:
WOMAC(Western Ontario and Mcmasters Universities) | Visit 2 (baseline) and Visit 3 (during the trial, 4week±7day) and Visit 4 (end of the trial) (12week±7day)
  The Western Ontario and McMaster Universities Arthritis Index (WOMAC) was assessed through a survey, with scores ranging from 0 to 96. Higher scores indicate worse outcomes.

SECONDARY OUTCOMES:
VAS(Visual Analogue Scale) | Visit 2 (baseline) and Visit 3 (during the trial, 4week±7day) and Visit 4 (end of the trial) (12week±7day)
  The Visual Analogue Scale (VAS) was assessed through a survey, with scores ranging from 0 to 100. Higher scores indicate worse outcomes.
Anti-inflammatory indicator | Visit 1 (screening) and Visit 3 (during the trial, 4week±7day) and Visit 4 (end of the trial) (12week±7day)
  Concentration of C-Reactive Protein (CRP) and Erythrocyte Sedimentation Rate (ESR) were measured from blood samples collected from the Jeonju vein after fasting for 8 hours and analyzed in our hospital's laboratory.

OTHER OUTCOMES:
Blood pressure | Visit 1 (screening) Visit 2 (baseline) and Visit 3 (during the trial, 4week±7day) and Visit 4 (end of the trial) (12week±7day)
  Blood pressure was measured in a sitting position after resting using BP-203 RVII(Colin Corp, Aichi, Japan).
Body weight | Visit 1 (screening)
  Body weight in kilograms were measured using a digital scale and stadiometer (BSM370, Biospace Co Ltd, Seoul).
Height | Visit 1 (screening)
  Height in meters were measured using a digital scale and stadiometer (BSM370, Biospace Co Ltd, Seoul).
Gathering subject information from the survey | Visit 1 (screening)
  All participants received information on demographics, history (diagnosis or drug treatment of hypertension, diabetes or dyslipidemia), health-related habits (smoking, drinking and alcohol), and medications taken through the survey. Participants were defined as non-smokers, past smokers, and current smokers, and non-smokers (0 to 98 g/week) or drinkers who drink an average of 7 cups of men and 5 or more cups of women twice per person.
Assessment of Bilateral Knee Joint Degeneration using AP/LAT Radiographs | Visit 1 (screening)
  Assessment of Bilateral Knee Joint Degeneration using AP/LAT Radiographs: Radiographic evaluation of bilateral knee joints will be performed using anterior-posterior (AP) and lateral (LAT) views. X-ray equipment in the hospital will be used to obtain these images. The degree of joint degeneration will be measured and reported based on established radiographic criteria, including the Kellgren-Lawrence grading scale.
Presence of Hepatitis B Surface Antigen (HbsAg) | Visit 1 (screening)
  At Visit 1, the presence of Hepatitis B Surface Antigen (HbsAg) was tested through blood analysis.
Presence of Hepatitis C Virus Antibodies (Anti-HCV) | Visit 1 (screening)
  At Visit 1, the presence of Hepatitis C Virus Antibodies (Anti-HCV) was tested through blood analysis.
Presence of Human Chorionic Gonadotropin (HCG) in Urine | Visit 1 (screening)
  At Visit 1, the presence of HCG in urine was tested for all females of reproductive age, excluding males and postmenopausal women.
Blood Glucose Level | Visit 1 (screening) and Visit 3 (during the trial, 4week±7day) Visit 4 (end of the trial) (12week±7day)
  Blood glucose level was measured from blood samples (12 cc) collected after fasting for 8 hours.
Complete Blood Count (CBC) | Visit 1 (screening) and Visit 3 (during the trial, 4week±7day) Visit 4 (end of the trial) (12week±7day)
  CBC was analyzed from blood samples (12 cc) collected after fasting for 8 hours.
Blood Urea Nitrogen (BUN) Level | Visit 1 (screening) and Visit 3 (during the trial, 4week±7day) Visit 4 (end of the trial) (12week±7day)
  BUN level was measured from blood samples (12 cc) collected after fasting for 8 hours.
Serum Creatinine Level | Visit 1 (screening) and Visit 3 (during the trial, 4week±7day) Visit 4 (end of the trial) (12week±7day)
  Serum creatinine level was measured from blood samples (12 cc) collected after fasting for 8 hours.
Estimated Glomerular Filtration Rate (GFR) | Visit 1 (screening) and Visit 3 (during the trial, 4week±7day) Visit 4 (end of the trial) (12week±7day)
  GFR was estimated from blood samples (12 cc) collected after fasting for 8 hours.
Total Cholesterol Level | Visit 1 (screening) and Visit 3 (during the trial, 4week±7day) Visit 4 (end of the trial) (12week±7day)
  Total cholesterol level was measured from blood samples (12 cc) collected after fasting for 8 hours.
Urine pH | Visit 1 (screening)
  The pH level of urine was measured at Visit 1 (screening) using a dipstick method.
Urine Specific Gravity | Visit 1 (screening)
  The specific gravity of urine was measured at Visit 1 (screening) using a refractometer.
Urine Protein | Visit 1 (screening)
  The protein level in urine was measured at Visit 1 (screening) using a dipstick method.
Urine Glucose | Visit 1 (screening)
  The glucose level in urine was measured at Visit 1 (screening) using a dipstick method.
Urine Ketones | Visit 1 (screening)
  The ketone level in urine was measured at Visit 1 (screening) using a dipstick method.
Urine Blood | Visit 1 (screening)
  The presence of blood in urine was measured at Visit 1 (screening) using a dipstick method.
Urine Leukocytes | Visit 1 (screening)
  The presence of leukocytes in urine was measured at Visit 1 (screening) using a dipstick method.
Aspartate Aminotransferase (AST) | Visit 1 (screening), Visit 3 (during the trial, 4 weeks ±7 days), Visit 4 (end of the trial, 12 weeks ±7 days)
  Aspartate Aminotransferase (AST) levels were measured using blood samples (12 cc) collected after fasting for 8 hours.
Alanine Aminotransferase (ALT) | Visit 1 (screening), Visit 3 (during the trial, 4 weeks ±7 days), Visit 4 (end of the trial, 12 weeks ±7 days)
  Alanine Aminotransferase (ALT) levels were measured using blood samples (12 cc) collected after fasting for 8 hours.
Alkaline Phosphatase (ALP) | Visit 1 (screening), Visit 3 (during the trial, 4 weeks ±7 days), Visit 4 (end of the trial, 12 weeks ±7 days)
  Alkaline Phosphatase (ALP) levels were measured using blood samples (12 cc) collected after fasting for 8 hours.
Gamma-Glutamyl Transferase (GGT) | Visit 1 (screening), Visit 3 (during the trial, 4 weeks ±7 days), Visit 4 (end of the trial, 12 weeks ±7 days)
  Gamma-Glutamyl Transferase (GGT) levels were measured using blood samples (12 cc) collected after fasting for 8 hours.
Total Bilirubin | Visit 1 (screening), Visit 3 (during the trial, 4 weeks ±7 days), Visit 4 (end of the trial, 12 weeks ±7 days)
  Total Bilirubin levels were measured using blood samples (12 cc) collected after fasting for 8 hours.
Serum Sodium (Na) | Visit 1 (screening), Visit 3 (during the trial, 4 weeks ±7 days), Visit 4 (end of the trial, 12 weeks ±7 days)
  Serum Sodium (Na) levels were measured from blood samples (12 cc) collected after fasting for 8 hours.
Serum Potassium (K) | Visit 1 (screening), Visit 3 (during the trial, 4 weeks ±7 days), Visit 4 (end of the trial, 12 weeks ±7 days)
  Serum Potassium (K) levels were measured from blood samples (12 cc) collected after fasting for 8 hours.
Serum Chloride (Cl) | Visit 1 (screening), Visit 3 (during the trial, 4 weeks ±7 days), Visit 4 (end of the trial, 12 weeks ±7 days)
  Serum Chloride (Cl) levels were measured from blood samples (12 cc) collected after fasting for 8 hours.
C-Reactive Protein (CRP) | Visit 1 (screening), Visit 3 (during the trial, 4 weeks ±7 days), Visit 4 (end of the trial, 12 weeks ±7 days)
  C-Reactive Protein (CRP) levels were measured from blood samples (12 cc) collected after fasting for 8 hours.
Erythrocyte Sedimentation Rate (ESR) | Visit 1 (screening), Visit 3 (during the trial, 4 weeks ±7 days), Visit 4 (end of the trial, 12 weeks ±7 days)
  Erythrocyte Sedimentation Rate (ESR) levels were measured from blood samples (12 cc) collected after fasting for 8 hours.
Triglycerides | Visit 1 (screening), Visit 3 (during the trial, 4 weeks ±7 days), Visit 4 (end of the trial, 12 weeks ±7 days)
  Triglyceride levels were analyzed from blood samples (12 cc) collected after fasting for 8 hours.
High-Density Lipoprotein (HDL) | Visit 1 (screening), Visit 3 (during the trial, 4 weeks ±7 days), Visit 4 (end of the trial, 12 weeks ±7 days)
  HDL levels were analyzed from blood samples (12 cc) collected after fasting for 8 hours.
Low-Density Lipoprotein (LDL) | Visit 1 (screening), Visit 3 (during the trial, 4 weeks ±7 days), Visit 4 (end of the trial, 12 weeks ±7 days)
  LDL levels were analyzed from blood samples (12 cc) collected after fasting for 8 hours.

CONTACTS AND LOCATIONS:
Locations (1):
- Pusan National University Hospital, Busan, Seo-gu, South Korea